CLINICAL TRIAL: NCT05676450
Title: Feasibility and Clinical Utility of Cell-free DNA (cfDNA) in Identifying Actionable Alterations and Minimal Residual Disease for Lymphoma Patients Across Community Centers in Texas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0603; NCI-2022-10562 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-15; First posted 2023-01-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Noninvasive Prenatal Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cell-free DNA (cfDNA) samples (Other): cell-free DNA (cfDNA) samples from DLBCL participants before and after treatment. cfDNA is DNA traveling in your blood outside of a cell and is easily collected from blood samples drawn using the vein puncture method.
  Blood will be drawn 3 times (by vein)
  Interventions: Diagnostic Test: cell-free DNA

INTERVENTIONS:
Diagnostic Test: cell-free DNA — Given by IV (vein)

SUMMARY:
To test the feasibility of collecting cell-free DNA (cfDNA) samples from DLBCL patients before and after treatment. cfDNA is DNA traveling in your blood outside of a cell and is easily collected from blood samples drawn using the vein puncture method.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the feasibility and clinical utility of ctDNA in identifying actionable alterations and minimal residual disease for lymphoma patients across community centers in Texas.

Secondary Objectives:

* To provide useful prognostic information before treatment, assess molecular response at interim time points and residual disease at the end of therapy, and identify tumor-specific mutations
* Levels of cfDNA and its association with both EFS and OS in patients receiving therapy

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients who are at least 18 years of age on the day of informed consent signing.
2. Patients must have a histologically documented diffuse large B-cell lymphoma requiring therapy.
3. Provision of written informed consent for the study.
4. Pregnant women not included
5. Cognitively impaired adults are not included.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | through study completion; an average 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chijioke Nze, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org